CLINICAL TRIAL: NCT04286646
Title: Correlation of Pupillary Diameter Change With Age and Anterior Chamber Depth After Cataract Surgery
Brief Title: Correlation of Pupillary Diameter Changewith Age and Anterior Chamber Depth After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Clinica Oftalmologica TACIR (Other)
Responsible Party: Principal Investigator, Enrique Ordiñaga-Monreal, OD, MSc, Clinical Optometrist, Clinica Oftalmologica TACIR
Other Study IDs: EC022018; 47/2018 (Other: CEIm Grupo Hospitalario Quirónsalud-Catalunya)
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Pupillary Disorders
Keywords: Cataract; Pupillary changes; Age; Anterior chamber depth
MeSH Terms: conditions — Pupil Disorders; Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pupil diameter before/after cataract: The investigators measure the pupil diameter before and after (3 months) cataract. Mesopic and photopic conditions

SUMMARY:
PURPOSE: To assess the correlation between the change in pupil diameter, age and depth of the anterior chamber after 3 months of cataract surgery both in photopic and mesopic conditions. And study the changes of the pupillary diameter at 3 months after surgery in the two light conditions

DETAILED DESCRIPTION:
Healthy patients who are going to be operated on for cataracts are expected to take part in the study. If during the clinical study the minimum number of patients established in the protocol is exceeded, new samples will continue to be registered until the end of the established period.

The sample selection mechanism is by consecutive recruitment during the study period (in order of arrival at the medical office). Patients are operated bilaterally in a period not exceeding 15 days and it will get the variables of both eyes. A simple random sampling will be used for the choice of single eye data per patient.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes with age equal to or greater than 45 years
* Diagnosed cataract N1, C1, P1 or worse in some eye.
* Patients who will be operated on both eyes.
* Patients who have not been diagnosed with diabetes mellitus.
* Patients who have given their informed consent to take part in the study.

Exclusion Criteria:

* Age under 45 years.
* Patients with anisocoria, neurological disorders, diagnosed with diabetes mellitus, glaucoma or another eye disease.
* Patients with complications during and after cataract surgery.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The field in which the study will be carried out is a private medical centre. TACIR Ophthalmology clinic is located in the TEKNON Medical Center in the city of Barcelona. The study population will be the patients of the TACIR ophthalmology clinic who will be operated on cataracts and agree to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Pupil diameter | Preoperatively and 3-months postoperatively
  It took measurements of pupil diameter in mesopic and photopic conditions using pupillometer software of the Topolyzer Vario (Wavelight Laser Technologie AG).
Anterior Chamber Depht | Preoperatively
  Anterior chamber depth was obtained with Pentacam® (Oculus Optikgeräte GmbH, Wetzlar, Germany).
Age | Preoperatively
  It took the patient's age at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ordiñaga-Monreal, OD, Principal Investigator — Clinica Oftalmologica TACIR
Locations (1):
- Clinica Oftalmológica TACIR, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanellopoulos AJ, Asimellis G, Georgiadou S. Digital pupillometry and centroid shift changes after cataract surgery. J Cataract Refract Surg. 2015 Feb;41(2):408-14. doi: 10.1016/j.jcrs.2014.05.049. PMID 25661135
- [Derived] Ordinaga-Monreal E, Castanera-Gratacos D, Castanera F, Fambuena-Muedra I, Vega F, Millan MS. Pupil size differences between female and male patients after cataract surgery. J Optom. 2022 Apr-Jun;15(2):179-185. doi: 10.1016/j.optom.2020.09.005. Epub 2021 Feb 3. PMID 33549502

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04286646/SAP_000.pdf
  • Informed Consent Form (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04286646/ICF_001.pdf